CLINICAL TRIAL: NCT00824928
Title: A Prospective Multicenter Registry of Salvage Cryotherapy in Recurrent Prostate Cancer Study
Brief Title: Salvage Cryotherapy in Recurrent Prostate Cancer
Acronym: SCORE
Status: Terminated | Type: Observational
Why Stopped: Study was ended due to low enrollment
Sponsor: University of Colorado, Denver (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 06-1040
Record Dates: First submitted 2009-01-15; First posted 2009-01-19 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2010-06

CONDITIONS: Recurrent Prostate Cancer
Keywords: Prostate Cancer; Recurrent Prostate Cancer; Prostate Cancer Recurrence; Radiation Failure; Salvage Cryotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cryosurgery; Cryotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Patients with locally recurrent prostate cancer that have chosen salvage cryotherapy
  Interventions: Procedure: Cryoablation / Cryotherapy

INTERVENTIONS:
Procedure: Cryoablation / Cryotherapy — Salvage Cryoablation of the prostate

SUMMARY:
To provide a systemic, uniform and user-friendly tool for collection of data on prostate cancer salvage cryotherapy in a multicenter setting. The goal is to learn more about the short and long term efficacy and safety of this procedure. Ultimately the data analysis will serve as a robust guidance instrument for improving upon the utilization of this procedure for the treatment of patients with recurrent (LRD) prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Read & understand informed consent related to this study including consenting and HIPPA authorization
* Undergone salvage cryotherapy of the prostate for recurrent prostate cancer

Exclusion Criteria:

* Patients who underwent radical prostatectomy as their primary therapy or other significant surgery (except prostatic biopsy)
* Patients with clinically confirmed distant metastasis (unless deemed beneficial by the treating physician)
* Any previous major rectal surgery
* Clinically significant lower urinary tract or rectal anomalies
* Existing urethral, rectal, or bladder fistulae

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Academic Institutions and Community Urologic Oncology Clinics in the United States of America and the United Kingdom
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2007-01; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Biochemical failure after treatment (defined as nadir PSA value + 2 ng/dl documented in the postoperative period). | 3-6 months intervals during the first 2 years after the completion of the procedure and yearly thereafter unless is amended by the treating physician

SECONDARY OUTCOMES:
Percentage change in QoL scores (EPIC) if available | 3-6 months intervals during the first 2 years after the completion of the procedure and yearly thereafter unless is amended by the treating physician
Percentage change in AUA-symptom score (also referred to as IPSS score) | 3-6 months intervals during the first 2 years after the completion of the procedure and yearly thereafter unless is amended by the treating physician
Percentage change in erectile dysfunction as measured by Sexual Health Inventory for men score (SHIM also referred to as IIEF score) | 3-6 months intervals during the first 2 years after the completion of the procedure and yearly thereafter unless is amended by the treating physician
Percentage change in urinary symptoms (continence score) | 3-6 months intervals during the first 2 years after the completion of the procedure and yearly thereafter unless is amended by the treating physician

CONTACTS AND LOCATIONS:
Overall Officials: Al Barqawi, MD, Study Chair — University of Colorado, Denver; David Crawford, MD, Study Chair — University of Colorado, Denver
Locations (17):
- United States (17):
  - Loma Linda University, Loma Linda, California
  - Kaiser Permanente, Sacremento, California
  - Prostate Institute of America, Ventura, California
  - University of Colorado at Denver and Health Sciences Center, Aurora, Colorado
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Midwest Urology/RMD Clinical Research, Melrose Park, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Methodist Hospital, Brooklyn, New York
  - Nelson Stone (private practice), New York, New York
  - Riverside Urology, Inc., Columbus, Ohio
  - Rhode Island Hospital/Warren Alpert Medical School of Brown University, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Cancer Institute - Memphis, Memphis, Tennessee
  - Urology Associates of North Texas, Arlington, Texas
  - Urology of Virginia, Sentara Medical Group, Norfolk, Virginia

REFERENCES:
- See also: Related Info — http://www.scorestudy.org